CLINICAL TRIAL: NCT03680950
Title: Efficacy Test of Real-Time Upper Gastrointestinal Monitoring System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: B-BR-106-096
Record Dates: First submitted 2018-09-17; First posted 2018-09-21 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-05

CONDITIONS: Upper Gastrointestinal Bleeding
MeSH Terms: conditions — Gastrointestinal Hemorrhage

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Upper Gastrointestinal Monitoring System (Experimental): Participants who meet criteria of enrollment and is willing to join in this study will wear a real-time upper gastrointestinal monitoring system for checking whether upper gastrointestinal rebleeding occurs continuously for 3 days.
  Interventions: Device: Upper Gastrointestinal Monitoring System

INTERVENTIONS:
Device: Upper Gastrointestinal Monitoring System — Participants will wear a monitoring system consisting of a tiny endoscopy and a mobile device. The endoscopy is inserted to upper gastrointestinal tract via nasal cavity and the mobile device is set to take and send images from the endoscopy to a server for analyzing if the abnormal condition occurs.

SUMMARY:
A monitoring system was developed for detecting upper gastrointestinal (UGI) rebleeding. This system consists of (1) a tiny endoscopy, (2) a wearable device, and (3) a software. The endoscopy is inserted to UGI tract via nasal cavity and then stayed there for 3 days. The wearable device is set to regularly receive the pictures from the endoscopy and sent to the software, which is able to automatically analyze whether the rebleeding occurs. This study aims to test the feasibility and efficacy of the monitoring system.

ELIGIBILITY:
Inclusion Criteria:

* "Rockall" score ≧3

Exclusion Criteria:

* Pregnant woman;
* Behavioral disorder;
* Major cognitive-perceptual deficit;
* The person who has a nasogastric (NG) tube;
* Other deficits or disorders that are not suitable for NG insertion;
* Participants who need to take MRI scan.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-10-12 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Time to detection of upper gastrointestinal rebleeding between the upper gastrointestinal monitoring system vs. the current monitoring index. | 3 days
  The real-time upper gastrointestinal monitoring system is compared with the current monitoring index. The efficacy is estimated by which monitoring method finding the upper gastrointestinal rebleeding first.

SECONDARY OUTCOMES:
The accuracy of upper gastrointestinal rebleeding detection between the upper gastrointestinal monitoring system vs. the current monitoring index. | 3 days
  The accuracy of the current monitoring index and the real-time upper gastrointestinal monitoring system is compared. The accuracy is estimated by calculating the ratio of the number of making false alarm and the number of finding re-bleeding right.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan